CLINICAL TRIAL: NCT00254800
Title: The Effect of Exenatide on Single and Multiple Doses Oral Contraceptive Pharmacokinetics in Healthy Female Subjects
Brief Title: The Effects of Exenatide on Oral Contraceptive Pharmacokinetics in Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H8O-EW-GWBC
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Ethinyl Estradiol; Levonorgestrel; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Experimental): Oral contraceptive 1 hour prior to exenatide/oral contraceptive 30 minutes after exenatide/oral contraceptive alone
  Interventions: Drug: ethinyl estradiol and levonorgestrel; exenatide
- Sequence 2 (Experimental): Oral contraceptive 30 minutes after exenatide/oral contraceptive alone/oral contraceptive 1 hour prior to exenatide
  Interventions: Drug: ethinyl estradiol and levonorgestrel; exenatide
- Sequence 3 (Experimental): Oral contraceptive alone/oral contraceptive 1 hour prior to exenatide/oral contraceptive 30 minutes after exenatide
  Interventions: Drug: ethinyl estradiol and levonorgestrel; exenatide

INTERVENTIONS:
Drug: ethinyl estradiol and levonorgestrel; exenatide — Oral contraceptive is ethinyl estradiol (30 μg) and levonorgestrel (150 μg) one time daily, per 28-day treatment period; Study drug (exenatide 10 mcg) is subcutaneously injected twice daily
  Other Names: Byetta; AC2993
  Arms: Sequence 1
Drug: ethinyl estradiol and levonorgestrel; exenatide — Oral contraceptive is ethinyl estradiol (30 μg) and levonorgestrel (150 μg) one time daily, per 28-day treatment period; Study drug (exenatide 10 mcg) is subcutaneously injected twice daily
  Other Names: Byetta; AC2993
  Arms: Sequence 2
Drug: ethinyl estradiol and levonorgestrel; exenatide — Oral contraceptive is ethinyl estradiol (30 μg) and levonorgestrel (150 μg) one time daily, per 28-day treatment period; Study drug (exenatide 10 mcg) is subcutaneously injected twice daily
  Other Names: Byetta; AC2993
  Arms: Sequence 3

SUMMARY:
The purpose of this study is the examine the effect of taking exenatide on the blood levels (pharmacokinetics) of orally-administered contraceptives.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal female of child-bearing potential.
* Body Mass Index (BMI) between 19 and 35 kg/m^2, inclusive.

Exclusion Criteria:

* On implanted contraceptives for 6 months, or injectable contraceptives for 12 months prior to the study.
* Evidence of diabetes mellitus.
* Participation in a study involving administration of an investigational compound within the past 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Assessment of Pharmacokinetics profile of exenatide measured by AUC and Cmax | Day 8 and Day 22 of each treatment period hours of sampling: Predose, 0.5, 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6,8, 10, 12, 16, 24, 48
  To evaluate the effect of exenatide on the multiple-dose pharmacokinetics of a combination oral contraceptive when administered one hour prior or 30 minutes after the exenatide dose.

SECONDARY OUTCOMES:
Assessment of Pharmacokinetics profile of exenatide measured by AUC and Cmax | Day 8 and Day 22 of each treatment period hours of sampling: Predose, 0.5, 1,1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6,8, 10, 12, 16, 24, 48
  To evaluate the effect of exenatide on the single-dose pharmacokinetics of the combination oral contraceptive when administered one hour prior or 30 minutes after the exenatide dose.
Safety and Tolerability assessment by Adverse events, clinical laboratory evaluations, vital signs, ECG blood glucose, body weight, physical examination and exenatide antibodies. | Baseline through Day 84
  Assessment of the safety and tolerability of concomitant administration of exenatide and the combination oral contraceptive by incidence of adverse events, Adverse events, clinical laboratory evaluations, vital signs, 12-lead electrocardiogram (ECG), blood glucose, body weight, physical examination and exenatide antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (1):
- Research Site, Plymouth, United Kingdom

REFERENCES:
- [Derived] Kothare PA, Seger ME, Northrup J, Mace K, Mitchell MI, Linnebjerg H. Effect of exenatide on the pharmacokinetics of a combination oral contraceptive in healthy women: an open-label, randomised, crossover trial. BMC Clin Pharmacol. 2012 Mar 19;12:8. doi: 10.1186/1472-6904-12-8. PMID 22429273